CLINICAL TRIAL: NCT05079464
Title: Exercise as a Primer for Excitatory Stimulation Study in Vascular Cognitive Impairment No Dementia (EXPRESS-V)
Brief Title: Exercise as a Primer for Brain Stimulation in Vascular Cognitive Impairment No Dementia (VCIND)
Acronym: EXPRESS-V
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3348
Record Dates: First submitted 2021-09-16; First posted 2021-10-15 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-11

CONDITIONS: Vascular Cognitive Impairment; Mild Cognitive Impairment
Keywords: transcranial direct current stimulation; tDCS; exercise; cognition; vascular cognitive impairment no dementia; vascular mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity | interventions — Transcranial Direct Current Stimulation; Exercise; Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized, blinded, repeated-session, parallel-design study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, outcomes assessors, and investigators will be blinded to stimulation type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise primed tDCS (Experimental): Individuals randomized to this group will receive exercise at University Health Network-Toronto Rehabilitation Institute followed by active tDCS.
  Interventions: Other: tDCS; Other: Exercise
- Exercise primed Sham stimulation (Other): Individuals randomized to this group will receive exercise at University Health Network-Toronto Rehabilitation Institute followed by sham tDCS.
  Interventions: Other: Exercise; Other: Sham stimulation
- Treatment as usual (exercise education) & tDCS (Other): Individuals randomized to this group will receive routine advice about physical activity, and active tDCS.
  Interventions: Other: tDCS; Other: Treatment as usual
- Treatment as usual (exercise education) & sham stimulation (Other): Individuals randomized to this group will receive routine advice about physical activity, and sham tDCS.
  Interventions: Other: Sham stimulation; Other: Treatment as usual

INTERVENTIONS:
Other: tDCS — All participants randomized to tDCS will receive active tDCS
  Arms: Exercise primed tDCS; Treatment as usual (exercise education) & tDCS
Other: Exercise — Participants will exercise at Toronto Rehab.
  Arms: Exercise primed Sham stimulation; Exercise primed tDCS
Other: Sham stimulation — The same procedure for tDCS will be used for the sham condition, except without active current.
  Arms: Exercise primed Sham stimulation; Treatment as usual (exercise education) & sham stimulation
Other: Treatment as usual — Exercise education/ treatment as usual will include routine advice about physical activity.
  Other Names: Exercise education
  Arms: Treatment as usual (exercise education) & sham stimulation; Treatment as usual (exercise education) & tDCS

SUMMARY:
People with vascular conditions are at risk of having memory problems, and these memory problems increase the risk for further cognitive decline. Brain stimulation has been used to improve mood and memory. Transcranial direct current stimulation (tDCS) is believed to work best on brain cells that are active or "primed" before stimulation. The purpose of this study is to compare the effects of exercise and tDCS on memory performance in patients who have completed cardiac rehabilitation and are at risk of cognitive decline.

DETAILED DESCRIPTION:
Vascular disease is a major risk factor and contributor to dementia. Current interventions to manage vascular risk factors have mixed results. Presently, there are no consistently effective treatments targeting vascular cognitive impairment no dementia.

Study Aim: To evaluate the effect of exercise-primed tDCS on global cognition.

Study Design: Eligible participants will be randomized to one of four interventions: Exercise primer with tDCS, Treatment as usual (TAU/exercise education) with tDCS, or Exercise primer with sham tDCS, Treatment as usual with sham tDCS. Participants randomized to an exercise group will undergo exercise, followed by either sham or active tDCS. Participants randomized to TAU will receive written information in accordance with the Canadian Physical Activity Guidelines for older adults and tDCS or sham. Cognition, behaviour, neuroimaging and blood biomarkers will be measured.

ELIGIBILITY:
Inclusion Criteria:

* ≥50 years of age; females must be post-menopausal
* Presence of cerebrovascular and/or cardiovascular risk factors or coronary artery disease
* Montreal Cognitive Assessment (MoCA) <27
* Sufficiently proficient in English
* Must be able to exercise at a moderate intensity level
* Presence of modest deficits (1 standard deviation below population norm) in one of the following domains: executive function, verbal memory, working memory, or visuospatial memory

Exclusion Criteria:

* History of stroke
* Change in psychotropics within the last 4 weeks
* Current benzodiazepine use due
* Metal implants that would preclude safe use of tDCS or neuroimaging
* Significant neurological or psychiatric conditions (current major depressive disorder, bipolar disorder, schizophrenia)
* MoCA <18 and/or clinical diagnosis of dementia
* Any medical contraindications to exercise

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment - Global Cognition | 2 weeks
  The Montreal Cognitive Assessment is a 5-minute test of global cognition and a validated tool for detecting early cognitive changes.

SECONDARY OUTCOMES:
Cognitive domains | 2 weeks
  Cognitive domains will be measured using the 60-minute battery recommended by the National Institute of Neurological Disorders and Stroke-Canadian Stroke Network.
Behavioural measures | 2 weeks
  Behaviour will be measured with the Mild Behavioural Impairment-Checklist.

CONTACTS AND LOCATIONS:
Overall Officials: Krista Lanctôt, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada